CLINICAL TRIAL: NCT00892996
Title: Efficacy of Prevention for Postoperative Nausea and Vomiting After Intrathecal Morphine in Cesarean Section: a Randomized Comparison of Metoclopramide or Ondansetron Alone or in the Combination With Dexamethasone.
Brief Title: Efficacy of Prevention for Postoperative Nausea and Vomiting After Intrathecal Morphine in Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Siriraj institutional review board, mahidol university
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Si 9091/2552(EC2)
Record Dates: First submitted 2009-05-03; First posted 2009-05-05 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Pregnancy; PONV
Keywords: Intrathecal morphine; Cesarean section; Nausea and vomiting; Prevention
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (No Intervention): Metoclopramide 10 mg intravenous
- 2 (No Intervention): Ondansetron 8 mg intravenous
- 3 (Active Comparator): dexamethasone 5 mg and metoclopramide 10 mg
  Interventions: Drug: dexamethasone
- 4 (Active Comparator): dexamethasone 5 mg and ondansetron 8 mg IV
  Interventions: Drug: dexamethasone 5 mg

INTERVENTIONS:
Drug: dexamethasone — Metoclopramide 10 mg and dexamethasone 5 mg intravenous
  Other Names: Dexamo
  Arms: 3
Drug: dexamethasone 5 mg — Ondansetron 8 mg and dexamethasone 5 mg IV
  Other Names: Dexamo
  Arms: 4

SUMMARY:
Post-operative nausea and vomiting are the major complications after spinal anesthesia with intrathecal morphine, therefore antiemetic drugs should be administered for best satisfaction of anesthesia to prevent these complication.

Furthermore, administration of a combination of antiemetic drugs with different mechanisms of action appears reasonable and synergistic effect of drugs.

In conclusion, we study efficacy of antiemetic effect of single antiemetic drug compare with combination antiemetic drugs.

DETAILED DESCRIPTION:
In this study : a randomized, double-blind, placebo-controlled, clinical trial comparing single doses of Metoclopramide 10 mg and Ondansetron 8 mg alone and a combination of Dexamethasone 5 mg and Metoclopramide 10 mg or a combination of Dexamethasone 5 mg and Ondansetron 8 mg for prevention of PONV after spinal morphine for cesarean section.

Inclusion criteria

1. Patient undergoes elective cesarean section age more than 18 years
2. Patient accepted in spinal anesthesia technique
3. ASA classification I-II
4. Patient understand question and evaluation process

Exclusion criteria

1. Hyperemesis gravidarum
2. Patient with ongoing antiemetic drugs treatment
3. Patient with history of drug allergy in Metoclopramide,Ondansetron and Dexamethasone

Outcome measurement By oral interview and nurse notification in 24 hr. post-operatively.

Detail of outcome measurement

1. Nausea and vomiting score
2. Pain score
3. Sedation score
4. Itch symptom
5. Patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy patients undergo Elective cesarean section age more than 18 years
* Patient accept spinal anesthesia technique
* ASA classification I-II
* Patient understand question and evaluation process

Exclusion criteria:

* Hyperemesis gravidarum
* Patient ongoing treatment with antiemetic drugs
* Allergy to Metoclopramide,Ondansetron and Dexamethasone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
nausea and vomiting after spinal anesthesia with intrathecal morphine in cesarean section | 24 hrs post operatively

SECONDARY OUTCOMES:
Secondary outcome measurement 1. Sedation score 2. Pain score 3. Itching symptom 4. Patient satisfaction | 24 Hrs post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Patchareya Nivatpumin, M.D., Principal Investigator — Anesthesiology department, Siriraj hospital, Mahidol University
Locations (1):
- Anesthesiology department, Siriraj hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Wu JI, Lo Y, Chia YY, Liu K, Fong WP, Yang LC, Tan PH. Prevention of postoperative nausea and vomiting after intrathecal morphine for Cesarean section: a randomized comparison of dexamethasone, droperidol, and a combination. Int J Obstet Anesth. 2007 Apr;16(2):122-7. doi: 10.1016/j.ijoa.2006.11.004. Epub 2007 Feb 1. PMID 17275282
- [Derived] Griffiths JD, Gyte GM, Popham PA, Williams K, Paranjothy S, Broughton HK, Brown HC, Thomas J. Interventions for preventing nausea and vomiting in women undergoing regional anaesthesia for caesarean section. Cochrane Database Syst Rev. 2021 May 18;5(5):CD007579. doi: 10.1002/14651858.CD007579.pub3. PMID 34002866